CLINICAL TRIAL: NCT05004792
Title: Correlation Between Online Case-based Training of Pathologists in Dermoscopic Images and Diagnostic Accuracy in Histopathological Interpretation of Skin Lesions Suspicious of Melanoma
Brief Title: Dermoscopy Augmented Histology Trial, a Randomized Controlled Trial
Acronym: DAHT-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Louisa Bønløkke Nervil, Medical doctor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AISC-DAHT, RCT
Record Dates: First submitted 2021-07-06; First posted 2021-08-13 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Melanoma; Pigmented Lesions
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial. Pathologists are randomized to either the control group or the intervention group, allocation ratio of 1:1.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participating Pathologists are either given access to a learning intervention called DermLoop Learn for a short period or not given access to any learning intervention. During the trial, both groups interpret histopathological skin lesions with access to clinical information, an overview picture, and a dermoscopic picture of the lesion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Access to DermLoop Learn IT platform
  Interventions: Other: DermLoop Learn
- Control group (No Intervention): No access to DermLoop Learn

INTERVENTIONS:
Other: DermLoop Learn — DermLoop Learn is our AI-augmented digital educational platform with case training on a library of 18,000+ benign and malignant skin lesions, educational videos on the correlation between dermoscopy and histology, as well as written learning modules for the most common skin lesion diagnosis. The education platform will give the user feedback on the image-based case training in dermoscopic diagnostic accuracy and adjust the cases depending on the user's progression.
  Arms: Intervention

SUMMARY:
Pathologists provide the current gold standard in skin lesion diagnostics, most often primarily based on the interpretation of histological slides. Still, it has been suggested that pathologists' diagnostic accuracy and confidence could be improved if they gained access to additional clinical information and in-vivo clinical and dermoscopic images of melanocytic tumors. This study examines the effect of digital training for pathologists in interpreting dermoscopic and clinical skin tumor images.

Aim:

To examine how case-based online training in interpreting clinical and dermoscopic images affects a pathologist's ability to diagnose skin tumors.

Data collection of DAHT cases: Department of plastic surgery, Herlev hospital, year 2020-2021,

DAHT platform: Made in 2021-2023 by Melatech,

Consensus agreement: Four dermatopathologists assess all DAHT cases, year 2023-2024

Enrollment of pathologists: Randomization and assessment DAHT cases, year 2025.

DETAILED DESCRIPTION:
Background Several publications suggest that the increasing melanoma incidence may partly be caused by histopathological overdiagnosis. Pathologists provide the current gold standard in skin lesion diagnostics, most often primarily based on the interpretation of histological slides. Still, it has been suggested that pathologists' diagnostic accuracy and confidence could be improved if they gained access to additional clinical information and in-vivo clinical and dermoscopic images of melanocytic tumors. However, it can be challenging to interpret clinical and dermoscopic images, and mastery typically requires more than six years of clinical experience. This learning journey can be significantly shortened if the trainee receives comprehensive training in pattern recognition for dermoscopy and clinical images, including immediate, accurate, and individualized feedback and access to a library with a large selection of skin lesion cases. This study examines the effect of digital training for pathologists in interpreting dermoscopic and clinical skin tumor images.

Former studies have only focused on melanocytic lesions. Still, most pathologists will receive both melanocytic and pigmented non-melanocytic lesions (seborrheic keratoses, dermatofibromas, etc.) due to clinical suspicion of melanoma. This study includes an un-filtered selection of 211 clinically melanoma-suspect skin lesions excised at a specialized surgical department; this material is named the DAHT cases.

Aim:

To examine how case-based online training in interpreting clinical and dermoscopic images affects a pathologist's ability to diagnose skin tumors.

Method Case Database

Lesion data were collected from patients between 02.11.2020 and 22.01.2021 at the Department of Plastic Surgery, Herlev Hospital. Requirements for eligibility for the current study are:

The patient was referred through the clinical cancer pathways for melanoma. The lesion was excised upon evaluation by the plastic surgeon.

Patients received oral and written information about the project and were asked to sign a consent form before participation. The participation did not affect the included patients' treatment, diagnostics, or follow-up. Upon consent, the following information was collected for each lesion:

Clinical image Dermoscopic image Patients´ CPR-number (personal ID-number) Sex and age of the patient Location of skin tumor (on a 3D avatar) Medical history (former treatment, congenital nevi, if pregnant, time of appearance of skin lesion, change in appearance, symptoms, former melanoma or other skin diseases, family history of melanoma, sun exposure within the last six months)

After excision, the specimen was prepared for pathological examination and a representative hematoxylin-eosin stain and, if available, a MelanA stain for each skin lesion was chosen for the study by an experienced dermatopathologist. These stains were subsequently digitized and coupled with the relevant information (dermoscopic and clinical image, tumor location, sex, age, lesion information, etc.). The CPR number was deleted, rendering the case anonymous. Each case is stored in a database under a random anonymous ID number.

Web-based IT platform

To maximize the number of pathologists that can be included in the study, the investigators have developed an IT platform for the trial (The DAHT platform). The platform enables the following features:

Sign-in Automated randomization Login Case presentation Diagnosis of cases and subquestions Tracking

The diagnostic options will be based on the standardized MPATH-Dx version 2.0 with additional non-melanocytic options based on the most common diagnoses to be excised due to suspicion of malignancy. After diagnosing the lesion, participating pathologists will rate their confidence and difficulty in the chosen diagnosis on a 6-step Likert scale similar to the one used in the MPATH-Dx system. They will also be asked whether they want a second opinion, if they need additional stains or tests, and which tests/stains. All cases will be presented in a randomized order unique to each participant.

The tracking feature will enable search pattern analysis, including time per diagnosis and percentage of time spent looking at the histology stain, dermoscopic image, clinical image, and clinical information.

Executive phase

General pathologists and dermatopathologists from Denmark, Australia, and other countries will be enrolled between 1.09.2023 and 1.12.2023. All participants will be sent an email informing them about the trial and the handling of their data before signing a digital consent. Upon inclusion, each enrolled pathologist will be asked to fill out a digital sign-in form with the following variables:

Name E-mail address (including verification) Age Sex Country Subspecialization (general pathologist or dermatopathologist) Number of years interpreting skin lesions Caseload from melanocytic lesions per month Percentage of caseload from melanocytic lesions Number of second opinion assessments per month Number of second opinion referrals per month Former training in dermoscopy (yes/no) Perceived relevance of dermoscopic images during histopathological evaluation on a 5-step Likert scale Routine with the use of digitized slides

Following the sign-in, all participants will be asked to answer a dermoscopy test consisting of 25 formerly validated test items. They will automatically be randomized (allocation ratio 1:1) to either the intervention or control group. Participants in the intervention group will receive immediate access to a previously developed digital (tablet or smartphone) educational platform for the dermoscopy of melanocytic lesions, watch educational videos on the correlation between dermoscopy and histology, and then answer the dermoscopy test again before diagnosing the lesions in this study. Participants in the control group will not be given access to the learning intervention but will diagnose the lesions from this study immediately after signing up and taking the dermoscopy test. Each participant will be asked to assess a minimum of 50 cases within 21 days, preferably all 211 cases.

Statistics:

The accuracy will be measured as the number of correct answers (validated by a former DAHT study: AISC-DAHT, consensus agreement) divided by the total number of answers. Inter-rater reliability will be measured using generalizability theory that allows calculations in nested and unbalanced designs. Mean time spent per diagnosis, perceived difficulty, and diagnostic confidence during the evaluation will be compared between the study groups using independent t-tests. A post hoc ANOVA will compare the time spent per diagnosis and the confidence of pathologists grouped by time spent training in dermoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologists are required to evaluate melanocytic lesions routinely
* Doctors must be registered authorized health personnel
* Access to a smartphone/tablet/computer with internet

Exclusion Criteria:

- Assessment of less than 50 DAHT cases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | 1 month
  Diagnostic accuracy according to specific diagnoses and sensitivity and specificity according to correct classification of malignant vs. benign lesions

SECONDARY OUTCOMES:
Inter-rater reliability | 1 month
  comparison of diagnosis between participants
time/case | 1 month
  Average time spent on each case
Average time spent on each image | 1 month
  Average time spent looking at the clinical image, dermoscopic image and histopathological image
use of clinical information | 1 month
  Whether the participants use the clinical information and when they decide to do so (before/after looking at the images)
Self-rated diagnostic confidence | 1 month
  participants average self-rated confidence on the cases
Perceived diagnostic difficulty | 1 month
  participants average perceived diagnostic difficulty on the cases
Dermoscopy test results | 1 month
  Difference between pre and post-dermoscopy tests
Second opinion | 1 month
  Number of requested second opinions and the underlying reason
Needs for stains | 1 month
  Needs for additional stains, including which stains
Needs for tests | 1 month
  Needs for additional tests (NGS, etc.), including which tests
training time vs time spent/DAHT case | 1 month
  Correlation between time spent training and time spent diagnosing DAHT cases.
MPATH-Dx specificity | 1 month
  Specificity according to MPATH-Dx classifications
MPATH-Dx sensitivity | 1 month
  Sensitivity according to MPATH-Dx classifications

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Bønløkke Nervil, Study Chair — Herlev Hospital, Denmark - Department of plastic surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glasziou PP, Jones MA, Pathirana T, Barratt AL, Bell KJ. Estimating the magnitude of cancer overdiagnosis in Australia. Med J Aust. 2020 Mar;212(4):163-168. doi: 10.5694/mja2.50455. Epub 2019 Dec 19. PMID 31858624
- [Background] Elmore JG, Barnhill RL, Elder DE, Longton GM, Pepe MS, Reisch LM, Carney PA, Titus LJ, Nelson HD, Onega T, Tosteson ANA, Weinstock MA, Knezevich SR, Piepkorn MW. Pathologists' diagnosis of invasive melanoma and melanocytic proliferations: observer accuracy and reproducibility study. BMJ. 2017 Jun 28;357:j2813. doi: 10.1136/bmj.j2813. PMID 28659278
- [Background] Scolyer RA, Soyer HP, Kelly JW, James C, McLean CA, Coventry BJ, Ferguson PM, Rawson RV, Mar VJ, de Menezes SL, Fishburn P, Stretch JR, Lee S, Thompson JF. Improving diagnostic accuracy for suspicious melanocytic skin lesions: New Australian melanoma clinical practice guidelines stress the importance of clinician/pathologist communication. Aust J Gen Pract. 2019 Jun;48(6):357-362. doi: 10.31128/AJGP-11-18-4759. PMID 31220881
- [Background] Ferrara G, Argenyi Z, Argenziano G, Cerio R, Cerroni L, Di Blasi A, Feudale EA, Giorgio CM, Massone C, Nappi O, Tomasini C, Urso C, Zalaudek I, Kittler H, Soyer HP. The influence of clinical information in the histopathologic diagnosis of melanocytic skin neoplasms. PLoS One. 2009;4(4):e5375. doi: 10.1371/journal.pone.0005375. Epub 2009 Apr 30. PMID 19404399
- [Background] Bedlow AJ, Cliff S, Melia J, Moss SM, Seyan R, Harland CC. Impact of skin cancer education on general practitioners' diagnostic skills. Clin Exp Dermatol. 2000 Mar;25(2):115-8. doi: 10.1046/j.1365-2230.2000.00590.x. PMID 10733633
- [Background] Badertscher N, Tandjung R, Senn O, Kofmehl R, Held U, Rosemann T, Hofbauer GF, Wensing M, Rossi PO, Braun RP. A multifaceted intervention: no increase in general practitioners' competence to diagnose skin cancer (minSKIN) - randomized controlled trial. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1493-9. doi: 10.1111/jdv.12886. Epub 2014 Dec 10. PMID 25491768
- [Background] Barnhill RL, Elder DE, Piepkorn MW, Knezevich SR, Reisch LM, Eguchi MM, Bastian BC, Blokx W, Bosenberg M, Busam KJ, Carr R, Cochran A, Cook MG, Duncan LM, Elenitsas R, de la Fouchardiere A, Gerami P, Johansson I, Ko J, Landman G, Lazar AJ, Lowe L, Massi D, Messina J, Mihic-Probst D, Parker DC, Schmidt B, Shea CR, Scolyer RA, Tetzlaff M, Xu X, Yeh I, Zembowicz A, Elmore JG. Revision of the Melanocytic Pathology Assessment Tool and Hierarchy for Diagnosis Classification Schema for Melanocytic Lesions: A Consensus Statement. JAMA Netw Open. 2023 Jan 3;6(1):e2250613. doi: 10.1001/jamanetworkopen.2022.50613. PMID 36630138
- [Result] Whiteman DC, Green AC, Olsen CM. The Growing Burden of Invasive Melanoma: Projections of Incidence Rates and Numbers of New Cases in Six Susceptible Populations through 2031. J Invest Dermatol. 2016 Jun;136(6):1161-1171. doi: 10.1016/j.jid.2016.01.035. Epub 2016 Feb 20. PMID 26902923
- [Result] Ternov NK, Vestergaard T, Holmich LR, Karmisholt K, Wagenblast AL, Klyver H, Hald M, Schollhammer L, Konge L, Chakera AH. Reliable test of clinicians' mastery in skin cancer diagnostics. Arch Dermatol Res. 2021 May;313(4):235-243. doi: 10.1007/s00403-020-02097-8. Epub 2020 Jun 28. PMID 32596742